CLINICAL TRIAL: NCT02561806
Title: A 52-Week Multicenter, Randomized, Blinded, Parallel-Group Study Comparing the Efficacy and Safety of Ixekizumab to Ustekinumab in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: IXORA-S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16012; I1F-MC-RHBS (Other: Eli Lilly and Company); 2015-000892-28 (EudraCT Number)
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ixekizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Ustekinumab (Active Comparator): 45 mg ustekinumab given as SC injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg at Week 0, 4, 16, 28, and 40. Placebo for ixekizumab injections will be used for blinding.
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Ixekizumab (Experimental): 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52.Placebo for ustekinumab injections will be used for blinding.
  Interventions: Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab
Drug: Ustekinumab — Administered SC
  Arms: Ustekinumab
Drug: Placebo — Administered SC

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug ixekizumab compared to ustekinumab in participants with moderate-to-severe-plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis for at least 6 months before baseline
* Failure, contraindication, or intolerability to at least 1 systemic therapy (including cyclosporine, methotrexate, or phototherapy)
* Psoriasis Area Severity Index (PASI) score at least 10 at screening and at baseline
* Participant must agree to use reliable method of birth control during the study; women must continue using birth control for at least 15 weeks after stopping treatment

Exclusion Criteria:

* Predominant pattern of pustular, erythrodermic, and/or guttate forms of psoriasis
* History of drug-induced psoriasis
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks before baseline and during the study
* Have received systemic nonbiologic psoriasis therapy or phototherapy within 4 weeks of baseline, or have had topical psoriasis treatment within the 2 weeks of baseline
* Concurrent or recent use of any biologic agent within the following washout periods: etanercept <28 days; infliximab, adalimumab, or alefacept <60 days; golimumab <90 days; rituximab <12 months; or any other biologic agent <5 half-lives prior to baseline
* Have prior use of ustekinumab, or have any condition or contraindication to ustekinumab that would preclude the participant from participating in this protocol
* Have previously completed or withdrawn from this study, participated in any other study with ixekizumab, have participated in any study investigating other interleukin (IL)-17 or IL-12/23 antagonists, or have received treatment with other IL-17 or IL-12/23 antagonists
* Have had a live vaccination within 12 weeks of baseline, or intend to have a live vaccination during the course of the study or within 15 weeks of completing treatment in this study
* Have had a vaccination with Bacillus Calmette-Guérin (BCG) within 12 months of baseline or intend to have vaccination with BCG during the course of the study or within 12 months of completing treatment in this study
* Have a known allergy or hypersensitivity to latex
* Have had any major surgery within 8 weeks of baseline or will require such during the study
* Have active or history of malignant disease within 5 years prior to baseline
* Significant uncontrolled disorder
* Ongoing infection or serious infection within 12 weeks of baseline; serious bone or joint infection within 24 weeks of baseline
* Are women who are lactating or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wein, Austria
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Edmonton
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Mississauga
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., North Bay
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., St. John's
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Martigues
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt am Main
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Witten
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kecskemét
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen, Netherlands
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Switzerland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geneva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lausanne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salford

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Armstrong A, Gonzalez-Cantero A, Khattri S, Muzy G, Malatestinic WN, Lampropoulou A, Feely M, See SK, Mert C, Blauvelt A. Comparing Achievement of National Psoriasis Foundation Treatment Targets among Patients with Plaque Psoriasis Treated with Ixekizumab versus Other Biologics in Clinical and Real-World Studies. Dermatol Ther (Heidelb). 2024 Apr;14(4):933-952. doi: 10.1007/s13555-024-01136-w. Epub 2024 Mar 23. PMID 38521874
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Wasel N, Thaci D, French LE, Conrad C, Dutronc Y, Gallo G, Berggren L, Lacour JP. Ixekizumab and Ustekinumab Efficacy in Nail Psoriasis in Patients with Moderate-to-Severe Psoriasis: 52-Week Results from a Phase 3, Head-to-Head Study (IXORA-S). Dermatol Ther (Heidelb). 2020 Aug;10(4):663-670. doi: 10.1007/s13555-020-00383-x. Epub 2020 May 15. PMID 32415575
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Plaque Psoriasis — http://www.lillytrialguide.com/EN-us/studies/psoriasis/rhbs

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Induction period occurring from week 0 to week 12 followed by maintenance period occurring week 12 to week 52 followed by post-treatment follow-up period occurring from last treatment period visit (week 52) or Early termination visit, for a minimum of 12 weeks following that visit.
Groups:
- Ustekinumab: 45 milligram (mg) ustekinumab given as subcutaneous (SC) injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg at Week 0, 4, 16, 28, and 40. Placebo for ixekizumab injections was used for blinding.
- Ixekizumab: 160 mg ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52. Placebo for ustekinumab injections was used for blinding.
Period: Induction Period
Arm/Group | Ustekinumab | Ixekizumab
Started | 166 | 136
Received At Least One Dose of Study Drug | 166 | 135
Completed | 164 | 131
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Site staff became unblinded | 1 | 0
Not completed — Randomized but not treated | 0 | 1
Period: Maintenance Period
Arm/Group | Ustekinumab | Ixekizumab
Started | 164 | 131
Completed | 151 | 123
Not Completed | 13 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Site staff became unblinded | 0 | 1
Period: Post-Treatment Follow-up
Arm/Group | Ustekinumab | Ixekizumab
Started | 157 (Participants who discontinued previous periods had option to enter post treatment follow-up period.) | 60 (Participants who discontinued previous periods had option to enter post treatment follow-up period.)
Completed | 155 | 59
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixekizumab: 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52. Placebo for ustekinumab injections will be used for blinding.
- Total: Total of all reporting groups
Arm/Group | Ustekinumab | Ixekizumab | Total
Number analyzed (Participants) | 166 | 136 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (13.25) | 42.7 (12.67) | 43.4 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 46 | 100
  Male | 112 | 90 | 202
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 157 | 125 | 282
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 12 | 11 | 23
  United Kingdom | 4 | 2 | 6
  Switzerland | 6 | 5 | 11
  Spain | 13 | 12 | 25
  Canada | 27 | 25 | 52
  Austria | 6 | 6 | 12
  Netherlands | 0 | 1 | 1
  Sweden | 4 | 2 | 6
  Belgium | 4 | 2 | 6
  Poland | 21 | 17 | 38
  Italy | 4 | 4 | 8
  France | 25 | 23 | 48
  Germany | 40 | 26 | 66
Weight [Mean (Standard Deviation); unit: Kilogram] | 89.4 (24.5) | 85.8 (20.30) | 87.8 (22.90)
Weight Categorical [Count of Participants; unit: Participants] — Population: All randomized participants who had baseline data.
  Participants
    <= 100 kg: number analyzed (Participants) | 166 | 135 | 301
    <= 100 kg | 121 | 104 | 225
    > 100 kg: number analyzed (Participants) | 166 | 135 | 301
    > 100 kg | 45 | 31 | 76
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: All randomized participants who had baseline data.
  kg/m^2
    number analyzed (Participants) | 166 | 135 | 301
    (all) | 29.7 (6.97) | 28.8 (5.55) | 29.3 (6.38)
Duration of psoriasis [Mean (Standard Deviation); unit: years] | 18.2 (12.0) | 18.0 (11.14) | 18.1 (11.60)
Age group at psoriasis onset [Count of Participants; unit: Participants]
  <40 years (Type 1 psoriasis) | 134 | 113 | 247
  >=40 years (Type 2 psoriasis) | 32 | 23 | 55
Psoriasis Area & Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, & legs). For each region the % area of skin involved was estimated from 0(0%) to 6(90%-100%) & severity was estimated by clinical signs of erythema, induration & scaling with scores range from 0 to 4 ("no" to "severe" involvement). Each area is scored & scores were combined for final PASI (sum of severity parameters for each region * area score * weighing factor [head(0.1), upper limbs(0.2), trunk(0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (most severe disease).
  units on a scale | 19.8 (9.02) | 19.9 (8.15) | 19.9 (8.62)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90) From Baseline
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for PASI 90. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Groups:
- Ustekinumab: 45 mg ustekinumab given as SC injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg at Week 0, 4, 16, 28, and 40. Placebo for ixekizumab injections was used for blinding.
- Ixekizumab: 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52. Placebo for ustekinumab injections was used for blinding.
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 136
percentage of participants | 42.2 | 72.8
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Non-Inferiority — Non-inferiority margin was -12.6% for 97.5% confidence interval; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.321, 97.5% CI 2-sided [0.198 to 0.445]

2. Secondary Outcome: Percentage of Participants With a ≥75% Improvement in PASI (PASI 75) From Baseline
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for PASI 75. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 136
percentage of participants | 68.7 | 88.2
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Ratio (RR) = 1.285, 95% CI 2-sided [1.130 to 1.439]

3. Secondary Outcome: Percentage of Participants With a 100% Improvement of PASI (PASI 100) From Baseline
Description: as for outcome 1
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for PASI 100. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Groups:
- Ustekinumab: 45 mg ustekinumab given as SC injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg at Week 0, 4, 16, 28, and 40. Placebo for ixekizumab injection was used for blinding.
- Ixekizumab: 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52. Placebo for ustekinumab injection was used for blinding.
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 136
percentage of participants | 14.5 | 36
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Superiority; p = 0.009, Regression, Logistic; Risk Ratio (RR) = 2.699, 95% CI 2-sided [1.423 to 3.975]

4. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1) With at Least a 2-Point Improvement From Baseline
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 12
Population: All randomized participants with baseline sPGA >=3 & received at least 1 dose of study drug and had a post-baseline measurement for sPGA. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 134
percentage of participants | 57.2 | 83.6
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Ratio (RR) = 1.469, 95% CI 2-sided [1.244 to 1.695]

5. Secondary Outcome: Percentage of Participants With a sPGA (0) Remission
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA assessed as 0, indicates complete resolution of plaque Ps.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for sPGA (0). Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 136
percentage of participants | 18.1 | 41.9
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Superiority; p = 0.021, Regression, Logistic; Risk Ratio (RR) = 3.421, 95% CI 2-sided [1.353 to 5.488]

6. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Psoriasis
Description: The percentage involvement of psoriasis on each participant's body surface area was assessed by the investigator on a scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand including palm, fingers and thumb.
  ANCOVA model with modified baseline observation carried forward (mBOCF) was used to produce Least Square (LS) mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug & had a baseline & post-baseline measurement for BSA affected by Ps.
  mBOCF: Participants who discontinued treatment due to Adverse Event (AE) were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Body Surface Affected
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 164 | 135
Percent Body Surface Affected | -16.92 [-18.50 to -15.34] | -22.55 [-24.34 to -20.76]

7. Secondary Outcome: Change From Baseline in Palmoplantar Psoriasis Severity Index (PPASI) Total Score
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 (no Ps) to 72. (the most severe disease) The PPASI was only assessed if participants have palmoplantar psoriasis at baseline.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants(Pts) who had psoriasis in palmoplantar regions at baseline & received at least 1 dose of study drug & had baseline & post-baseline PPASI data.
  mBOCF:Pts who discontinued treatment due to AE were imputed by their baseline observation, Pts who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 28 | 35
units on a scale | -8.34 [-9.64 to -7.03] | -10.31 [-11.63 to -8.99]

8. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI) Total Score
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had psoriasis in scalp region at baseline & received at least 1 dose of study drug & had baseline & post-baseline PSSI data.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 152 | 119
units on a scale | -16.00 [-17.24 to -14.77] | -19.29 [-20.67 to -17.92]

9. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Total Score
Description: NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail(fn) Ps. This scale is used to evaluate severity of fn bed Ps & fn matrix Ps by area of involvement in the fn unit. fn is divided with imaginary horizontal & longitudinal lines into quadrants. Each fn is given a score for fn bed Ps 0(none) to 4(Ps in 4 quadrants of the fn) & fn matrix Ps 0(none) to 4(Ps in 4 quadrants in matrix), depending on presence (score of 1) or absence (score of 0) of any of the features of fn bed or matrix Ps in each quadrant.NAPSI score of a fn is sum of scores in fn bed & fn matrix from each quadrant (maximum of 8). Each fn is evaluated, then the sum of all fn equals the total NAPSI score with a range from range 0 to 80. Higher scores indicate more severe ps.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had nail psoriasis at baseline & received at least 1 dose of study drug and had baseline & post-baseline NAPSI measurement.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 103 | 84
units on a scale | -5.02 [-7.19 to -2.84] | -12.24 [-14.72 to -9.77]

10. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for Itch NRS.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 165 | 135
units on a scale | -4.12 [-4.51 to -3.74] | -4.56 [-4.98 to -4.14]

11. Secondary Outcome: Change From Baseline on the Skin Pain Visual Analog Scale (VAS) (0,100)
Description: Skin Pain VAS is a participant administered scale designed to measure skin pain from psoriasis using a 100-millimeter (mm) horizontal VAS. Overall severity of a participant's skin pain from psoriasis at the present time is indicated by placing a single mark on the horizontal scale (0 = no skin pain; 100 = severe skin pain).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for skin pain VAS.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 165 | 135
mm | -29.92 [-32.81 to -27.04] | -33.32 [-36.44 to -30.20]

12. Secondary Outcome: Percentage of Participants With Dermatology Life Quality Index (DLQI) (0,1)
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment). A score of 0 or 1 indicates no impact of disease on a participants quality of life.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for DLQI. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 166 | 136
percentage of participants | 44.6 | 61.0
Statistical Analysis 1: Comparison: Ustekinumab vs Ixekizumab; Test type: Superiority; p = 0.012, Regression, Logistic; Risk Ratio (RR) = 1.391, 95% CI 2-sided [1.085 to 1.698]

13. Secondary Outcome: Change From Baseline on the Hospital Anxiety and Depression Scale (HADS) Depression Subscale
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 items questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for HADS depression subscale.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 162 | 134
units on a scale | -0.96 [-1.38 to -0.54] | -1.20 [-1.65 to -0.74]

14. Secondary Outcome: Change From Baseline on the Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale.
Description: as for outcome 13
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for HADS anxiety subscale.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 162 | 134
units on a scale | -0.90 [-1.37 to -0.43] | -1.27 [-1.80 to -0.73]

15. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score;
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. SF-36 acute version was used, which has a 1 week recall period.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for SF-36 PCS score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Ustekinumab: 45 mg ustekinumab given as SC injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg at Week 0, 4, 16, 28, and 40. Placebo for ixekizumab injection was be used for blinding.
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 164 | 133
units on a scale | 3.10 [1.97 to 4.23] | 5.03 [3.80 to 6.26]

16. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Mental Component Summary (MCS) Score
Description: as for outcome 15
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for SF36 MCS score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 164 | 133
units on a scale | 2.36 [0.87 to 3.86] | 2.96 [1.33 to 4.59]

17. Secondary Outcome: Change From Baseline on Patient Global Assessment of Disease Severity (PatGA)
Description: The Patient Global Assessment of Disease Severity is a single-item participant-reported outcome measure on which participants are asked to rate the severity of their psoriasis "today" from 0 (Clear) = no psoriasis, to 5 (Severe) = the worst their psoriasis has ever been.
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for PatGA.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 164 | 135
units on a scale | -2.60 [-2.78 to -2.42] | -3.07 [-3.26 to -2.88]

18. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D 5L) "Bolt On" Psoriasis (PSO) -Index
Description: The European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of a descriptive system of the respondent's health which comprises the following 5 dimensions: 1) mobility 2) self-care 3) usual activities 4) pain/discomfort 5) anxiety/depression. The Bolt On PSO is an addition to the EQ-5D-5L that consists of 2 dimensions specific to psoriatic disease: 6) skin irritation (itching) and 7) self-confidence. Index scores for the Bolt On PSO range from 0.0042 to 1.0 (worse to better health).
  ANCOVA model was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for EQ-5D 5L "Bolt On" PSO-Index.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 165 | 134
units on a scale | 0.11 [0.09 to 0.13] | 0.15 [0.13 to 0.17]

19. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D 5L) VAS
Description: The EQ-5D 5L is a standardized measure of health status that includes a descriptive system of the respondent's health and a rating of his/her current health state using a 0 (worst health imaginable)- to 100 (best health imaginable)-millimeter (mm) Visual Analog Scale (VAS). ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for EQ-5D 5L VAS.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- Ixekizumab: 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg ixekizumab given as a single SC injection once every 2 weeks from week 2 through week 12. After week 12 participants will receive 80 mg ixekizumab every 4 weeks through week 52. Placebo for ustekinumab injectio was used for blinding.
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 163 | 134
mm | 8.75 [5.77 to 11.74] | 12.24 [9.01 to 15.46]

20. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D 5L) United Kingdom(UK) Population-based Index Score
Description: The EQ-5D-5L descriptive system comprises 5 dimensions, each with 5 levels. The EQ-5D-5L health states were converted into a single summary index by applying a crosswalk using a UK Population value set to each of the levels in each dimension. This produced patient-level index scores between -0.594 and 1.0 (worse to better health).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug & had baseline & post-baseline EQ-5D 5L UK population-based index score measurement.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 165 | 134
units on a scale | 0.12 [0.09 to 0.15] | 0.15 [0.12 to 0.18]

21. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Absenteeism
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work & WPAI-PSO absenteeism score is derived from these questions. Each WPAI score is expressed as an impairment percentage (0-100), with higher scores representing greater impairment (worse outcomes).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for WPAI-PSO absenteeism score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 90 | 87
units on a scale | -1.42 [-4.55 to 1.72] | -0.46 [-3.51 to 2.60]

22. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Presenteeism
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work & WPAI-PSO Presenteeism score is derived from these questions. each WPAI score is expressed as an impairment percentage (0-100), with higher scores representing greater impairment (worse outcomes).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for WPAI-PSO presenteeism score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 98 | 92
units on a scale | -15.53 [-18.33 to -12.72] | -16.91 [-19.71 to -14.11]

23. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Work Impairment Score.
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work & WPAI-PSO work impairment score is derived from these questions. each WPAI score is expressed as an impairment percentage (0-100), with higher scores representing greater impairment (worse outcomes).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for WPAI-PSO work impairment score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 90 | 87
units on a scale | -15.05 [-19.25 to -10.85] | -16.27 [-20.39 to -12.16]

24. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Impairment in Activities Performed Outside of Work
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work & WPAI-PSO impairment in activities performed outside of work score is derived from these questions. each WPAI score is expressed as an impairment percentage (0-100), with higher scores representing greater impairment (worse outcomes).
  ANCOVA model with mBOCF was used to produce LS mean with baseline, treatment group, region weight group as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants(Pts) who received at least 1 dose of study drug & had baseline & post-baseline data for WPAI-PSO impairment in activities performed outside work.
  mBOCF:Pts who discontinued treatment due to AE were imputed by their baseline observation, pts who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ustekinumab | Ixekizumab
Number analyzed (Participants) | 154 | 127
units on a scale | -19.14 [-21.79 to -16.48] | -23.06 [-26.04 to -20.09]

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose study drug.
Groups:
- Ustekinumab - Induction; Ustekinumab - Maintenance: 45 milligram (mg) Ustekinumab given as subcutaneous (SC) injection for participants ≤100 kilograms (kg) and 90 mg SC injection for participants >100 kg. Placebo for Ixekizumab injection was used for blinding.
- Ixekizumab - Induction: 160 mg Ixekizumab given as two subcutaneous (SC) injections at baseline followed by 80 mg Ixekizumab given as a single SC injection once every 2 weeks.
  Placebo for Ustekinumab injection was used for blinding.
- Ixekizumab - Maintenance: 80 mg Ixekizumab given as a single SC injection once every 4 weeks. Placebo for Ustekinumab injection was used for blinding.
- Ustekinumab - Post Treatment Follow up; Ixekizumab - Post Treatment Follow up: Participants were allowed to continue the treatment administered during the blinded period or any other psoriasis treatment.
Arm/Group | Ustekinumab - Induction | Ixekizumab - Induction | Ustekinumab - Maintenance | Ixekizumab - Maintenance | Ustekinumab - Post Treatment Follow up | Ixekizumab - Post Treatment Follow up
Serious Adverse Events (participants affected / at risk) | 0/166 | 2/135 | 6/164 | 7/131 | 2/157 | 0/60
Other Adverse Events (participants affected / at risk) | 55/166 | 40/135 | 65/164 | 50/131 | 0/157 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab - Induction (N=166) | Ixekizumab - Induction (N=135) | Ustekinumab - Maintenance (N=164) | Ixekizumab - Maintenance (N=131) | Ustekinumab - Post Treatment Follow up (N=157) | Ixekizumab - Post Treatment Follow up (N=60)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab - Induction (N=166) | Ixekizumab - Induction (N=135) | Ustekinumab - Maintenance (N=164) | Ixekizumab - Maintenance (N=131) | Ustekinumab - Post Treatment Follow up (N=157) | Ixekizumab - Post Treatment Follow up (N=60)
Injection site erythema (General disorders) | 0 (0) | 10 (15) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 34 (39) | 23 (27) | 40 (52) | 36 (47) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 11 (16) | 8 (8) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 9 (11) | 5 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (17) | 7 (9) | 12 (19) | 10 (17) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 11 (11) | 4 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days